CLINICAL TRIAL: NCT07348237
Title: An Open-Label, Single-Dose Clinical Study to Evaluate the Pharmacokinetics of MK-2828 in Participants With Renal Impairment
Brief Title: A Clinical Trial of MK-2828 in People With Kidney Disease (MK-2828-006)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2828-006; MK-2828-006 (Other: MSD)
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Failure; End-Stage Renal Disease; Renal Impairment
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Severe Renal Impairment (Experimental): Participants with severe renal impairment will receive a single dose of MK-2828 on Day 1
  Interventions: Drug: MK-2828
- End Stage Renal Disease (ESRD) on Hemodialysis (HD) (Experimental): Participants with ESRD will receive a single dose of MK-2828 on Day 1 in each of 2 periods, with a washout of at least 14 days between doses.
  Interventions: Drug: MK-2828
- Healthy Mean Matched Control (Experimental): Participants with normal renal function will receive a single dose of MK-2828 on Day 1
  Interventions: Drug: MK-2828

INTERVENTIONS:
Drug: MK-2828 — Oral administration

SUMMARY:
The goal of this trial is to measure what happens to 1 or 2 doses of MK-2828 in a person's body over time (pharmacokinetic or PK trial). Researchers want to learn if the PK of people with certain types of kidney disease is similar to the PK of healthy people.

ELIGIBILITY:
The main inclusion criteria include but are not limited to the following:

* Is in generally good health, with the exception of renal impairment participants. Participants with stable, chronic medical or psychiatric conditions may be included at the discretion of the investigator and the Sponsor.

Severe Renal Impairment Participants:

* Has an estimated glomerular filtration rate (eGFR) < 30 mL/min), but is not on hemodialysis (HD)

ESRD on HD Participants:

* Has ESRD maintained on stable outpatient regimen of intermittent high-flux HD at a healthcare center for > 3 months prior to study entry

The main exclusion criteria include but are not limited to the following:

Renal Impairment Participants:

* History of any illness, other than renal impairment, that, in the opinion of the investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study.

Healthy Matched Control Participants:

* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases. Participants with a remote history of uncomplicated medical events (eg, uncomplicated kidney stones, as defined as spontaneous passage and no recurrence in the last 5 years, or childhood asthma) may be enrolled in the study at the discretion of the investigator.

Ages: 24 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2026-08-18 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of MK-2828 in Plasma | Pre dose and at designated time points up to 192 hours post dose
  Blood samples will be collected to determine the AUC0-inf of MK-2828
Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-last) of MK-2828 in Plasma | Pre dose and at designated time points up to 192 hours post dose
  Blood samples will be collected to determine the AUC0-last of MK-2828
Area Under the Concentration-time Curve From Time 0 to 24 Hours Postdose (AUC0-24) of MK-2828 in Plasma | Pre dose and at designated time points up to 24 hours post dose
  Blood samples will be collected to determine the AUC0-24 of MK-2828
Maximum Plasma Concentration (Cmax) of MK-2828 in Plasma | Pre dose and at designated time points up to 192 hours post dose
  Blood samples will be collected to determine the Cmax of MK-2828
Time of the Maximum Observed Concentration (Tmax) of MK-2828 in Plasma | Pre dose and at designated time points up to 192 hours post dose
  Blood samples will be collected to determine the Tmax of MK-2828
Concentration at 24 Hours Postdose (C24) of MK-2828 in Plasma | At designated time points up to 24 hours post dose
  Blood samples will be collected to determine the C24 of MK-2828
Apparent Terminal Elimination Half-life (t1/2) of MK-2828 in Plasma | Pre dose and at designated time points up to 192 hours post dose
  Blood samples will be collected to determine the t1/2 of MK-2828
Apparent Total Plasma Clearance (CL/F) of MK-2828 | Pre dose and at designated time points up to 192 hours post dose
  Blood samples will be collected to determine the CL/F of MK-2828
Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) of MK-2828 in Plasma | Pre dose and at designated time points up to 192 hours post dose
  Blood samples will be collected to determine the Vz/F of MK-2828

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 14 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 2 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Area Under the Concentration-time Curve From Start to End of Dialysis (AUCD) of MK-2828 | Prior to hemodialysis (HD) and at designated time points until day 6
  Blood samples will be collected to determine the AUCD of MK-2828
Area Under the Concentration-time Curve Determined from the Pre-dialyzer Line (AUCCa) of MK-2828 | Prior to hemodialysis (HD) and at designated time points until day 6
  Blood samples will be collected to determine the during AUCCa of MK-2828 during the dialysis period
Area Under the Concentration-time Curve Determined from the Post-dialyzer Line (AUCCv) of MK-2828 | Prior to hemodialysis (HD) and at designated time points until day 6
  Blood samples will be collected to determine the during AUCCv of MK-2828 during the dialysis period
Dialysis Clearance (CLD) of MK-2828 Based on Plasma | Prior to hemodialysis (HD) and at designated time points until day 6
  Blood samples will be collected to determine the CLD of MK-2828 based on plasma during the dialysis period
Hemodialysis Extraction Ratio (ER_D) of MK-2828 | Prior to hemodialysis (HD) and at designated time points until day 6
  Blood samples will be collected to determine the ER_D of MK-2828 during the dialysis period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com